CLINICAL TRIAL: NCT00594802
Title: Systemic Reactions to Allergen Immunotherapy Amd Skin Testing
Acronym: chackos
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: DR. RICHARD F LOCKEY, UNIVERSITY OF SOUTH FLORIDA
Other Study IDs: systemic reaction protocol
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2008-07

CONDITIONS: SYSTEMIC REACTION
Keywords: ALLERGIC REACTION
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHART REVIEW ONLY: CHART REVIEW OF PATIENTS WITH SYSTEMIC REACTIONS

SUMMARY:
Allergy skin tests and allergen immunotherapy are common procedures for both the diagnosis and treatment of atopic diseases. Allergen immunotherapy has proved to be effective in reducing the symptoms of allergic rhinitis and asthma1-2. Despite its clinical benefit, there is risk of systemic reactions associated with these procedures.

The systemic reaction rate to skin testing for aeroallergens is significant lower than the rate of reactions to immunotherapy, but it is not negligible. Lin et al reported only 2 patients who had systemic allergic reactions to skin testing for respiratory allergies in 10,400 patients tested.3 They determined the overall risk of inducing anaphylactic reactions by skin testing to be less than 0.02% and other studies have produced similar results.4-5 The rate of systemic reactions to skin testing is likely underscored. Thompson et. al reported a systemic reaction rate of 6% of patients receiving skin testing.6 It is important to recognize the risk of systemic reactions seeing skin testing is commonly done. It is also imperative to recognize the treatments for these reactions to prevent progression.

Hypothesis The systemic reaction rate to allergen immunotherapy and skin testing to aeroallergens is higher than previously reported. Biphasic anaphylactic reactions rarely occur with allergen immunotherapy and skin testing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who are receiving skin testing or allergen immunotherapy from one allergy practice.

Exclusion Criteria:

* NON Male and female subjects who are receiving skin testing or allergen immunotherapy from one allergy practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects who are receiving skin testing or allergen immunotherapy from one allergy practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
This is a prospective observational study of patients who are having either skin testing or allergen immunotherapy for the diagnosis or treatment of allergic rhinitis, conjunctivitis, and/or asthma.

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD F LOCKEY, MD, Principal Investigator — USF DIRECTOR OF ALLERGY AND IMMUNOLOGY
Locations (1):
- USF, Tampa, Florida, United States

REFERENCES:
- [Derived] Bagg A, Chacko T, Lockey R. Reactions to prick and intradermal skin tests. Ann Allergy Asthma Immunol. 2009 May;102(5):400-2. doi: 10.1016/S1081-1206(10)60511-X. PMID 19492661